CLINICAL TRIAL: NCT05130762
Title: A Post-Market Clinical Follow Up Study to Evaluate BD PureHub™ Disinfecting Cap Use on Needle-Free Connectors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MDS-20PUREU001
Record Dates: First submitted 2021-10-08; First posted 2021-11-23 (Actual); Results first posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-03

CONDITIONS: Catheter Related Complication; Vascular Access Site Management; Disinfecting Cap

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- General Cohort (Other): All patients who receive a VAD as standard of care in combination with needle-free connectors. A BD PureHub™ Disinfecting Cap will be placed on each eligible needle-free connector and all attachments/removals incl. reason for change will be documented up to 45 days post-enrollment date.
  Interventions: Device: BD PureHub™ Disinfecting Cap Placements: Attachments/removals

INTERVENTIONS:
Device: BD PureHub™ Disinfecting Cap Placements: Attachments/removals — Attachment/Removals of BD PureHub™ Disinfecting Cap

SUMMARY:
The study will collect use data of the Becton Dickinson (BD) PureHub™ Disinfecting Cap in combination with needle-free connectors, which are attached to vascular access devices (VAD).

DETAILED DESCRIPTION:
This is a multi-center, prospective observational study of a minimum of 150 study participants who have vascular access devices (VADs) with needle-free connectors as part of their routine medical care.

Patients will be followed from the time of enrollment through the duration of VAD therapy or 45 days post enrollment date, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Has an eligible vascular access device with needle-free connectors in situ or will have one placed Note: This covers all needle-free devices, including central venous catheters, peripheral IV catheters and arterial VADs
2. Is expected to receive VAD therapy for a minimum of 3 days
3. Is expected to be available for regular observation from consent until end of study
4. Able and willing to provide informed consent or legal authorized representative (LAR) authorized to give consent on behalf of the participant

Exclusion Criteria:

1. BD PureHub™ Disinfecting Cap or any other disinfecting cap in place for more than twelve (12) hours (>12 hours) prior to study participation
2. Presence of any infection, bacteremia, or septicemia is known or suspected
3. Any condition which, in the opinion of the Investigator, precludes the participant from participation in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Medical University Vienna, Vienna, Austria
- UZA, Antwerp, Belgium
- Azienda Ospedaliera Universitaria Careggi, Florence, Italy
- Spain (2):
  - Hospital Universitario de A Coruña, A Coruña
  - Hospital Universitari Arnau de Vilanova, Valencia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | General Cohort
Started | 157
Completed | 156
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Enrolled: All participants who signed the ICF Evaluable : All enrolled participants who had at least 1 BD PureHub™ Disinfecting Cap applied.
Arm/Group | General Cohort
Number analyzed (Participants) | 157
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 78
  >=65 years | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (20.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77
  Male | 80
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 154
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Austria | 30
  Belgium | 14
  Italy | 48
  Spain | 65

OUTCOME MEASURES:

1. Primary Outcome: Attachment & Removal Success Rate of the BD PureHub Disinfecting Caps to a Needle-free Connector
Description: * Attachment success rate of the BD PureHub™ Disinfecting Caps to a needle-free connector (successful attachment/total number of attachments)
  * Removal success rate of the BD PureHub™ Disinfecting Caps to a needle-free connector (successful removal/ total number of intended removals)
Time Frame: Up to 45 days post-enrollment date
Population: The primary objective was to assess the rate of select performance measures (attachment success rate & removal success rate) of the BD PureHub™ Disinfecting Caps on swabbable NFC when used in a clinical environment.
Measure: Number (95% Confidence Interval); unit: percentage of attachment success rate
Groups:
- Attachment: All patients who receive a VAD as standard of care in combination with needle-free connectors. A BD PureHub™ Disinfecting Cap will be placed on each eligible needle-free connector and all attachments/removals incl. reason for change will be documented up to 45 days post-enrollment date.
  BD PureHub™ Disinfecting Cap Placements:Attachment of BD PureHub™ Disinfecting Cap
- Removals: All patients who receive a VAD as standard of care in combination with needle-free connectors. A BD PureHub™ Disinfecting Cap will be placed on each eligible needle-free connector and all attachments/removals incl. reason for change will be documented up to 45 days post-enrollment date.
  BD PureHub™ Disinfecting Cap Placements: Removals of BD PureHub™ Disinfecting Cap
Arm/Group | Attachment | Removals
Number analyzed (Participants) | 156 | 156
percentage of attachment success rate | 99.9 [99.6 to 100] | 99.7 [99.2 to 99.9]

2. Primary Outcome: Number of Participants With BD PureHub™ Disinfecting Cap Device-related Adverse Events.
Description: Rate of device-related adverse events
Time Frame: Up to 45 days post-enrollment date
Population: AEs in the Enrolled Population
Measure: Number; unit: participants
Arm/Group | General Cohort
Number analyzed (Participants) | 157
participants | 0

ADVERSE EVENTS:
Time Frame: Participants were followed from the time of enrollment until one week post VAD therapy, department/hospital discharge or 45 days post enrollment date, whichever came first.
Arm/Group | General Cohort
All-Cause Mortality (participants affected / at risk) | 2/157
Serious Adverse Events (participants affected / at risk) | 2/157
Other Adverse Events (participants affected / at risk) | 0/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | General Cohort (N=157)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — A 72-year-old male participant died as an aggravation of his oncological disease shortly after enrollment in the study.
Respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1) — a 77-year-old male participant who died due to respiratory insufficiency after a long chronical disease.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT05130762/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-08): https://cdn.clinicaltrials.gov/large-docs/62/NCT05130762/SAP_001.pdf